CLINICAL TRIAL: NCT01074060
Title: A Phase I/Pilot Study of Intravenous PLERIXAFOR Following Cyclophosphamide Mobilization in Patients With Multiple Myeloma
Brief Title: Plerixafor and Filgrastim Following Cyclophosphamide for Stem Cell Mobilization in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08186; NCI-2010-00160
Record Dates: First submitted 2010-02-19; First posted 2010-02-24 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — plerixafor; Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): MOBILIZATION: Patients receive cyclophosphamide IV. Patients also receive filgrastim subcutaneously (SC) daily beginning approximately 24 hours later.
  TREATMENT/APHERESIS: Beginning 10 days after cyclophosphamide, patients receive plerixafor IV over 30 minutes followed by filgrastim SC on each day of apheresis.
  Interventions: Drug: plerixafor; Biological: filgrastim; Drug: cyclophosphamide; Procedure: autologous hematopoietic stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: plerixafor — Given IV
  Other Names: AMD 3100; LM-3100; Mozobil
Biological: filgrastim — Given SC
  Other Names: G-CSF; granulocyte colony-stimulating factor; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Procedure: autologous hematopoietic stem cell transplantation — autologous hematopoietic stem cell transplantation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: There are different methods of stem cell mobilization, such as using colony-stimulating factors alone or following chemotherapy priming. More recently, the combination of plerixafor and colony-stimulating factors has been shown to enhance stem cell mobilization. This study will assess whether the combination of plerixafor and Granulocyte Colony-Stimulating Factor (G-CSF) is effective following chemotherapy mobilization with cyclophosphamide.

PURPOSE: To assess the safety, tolerability, and best dose of intravenous plerixafor following cyclophosphamide priming.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of intravenous(IV) PLERIXAFOR when given in combination with cyclophosphamide and G-CSF as a mobilization regimen in patients with Multiple Myeloma.

SECONDARY OBJECTIVES:

I. To determine if intravenous PLERIXAFOR, given with a cyclophosphamide and G-CSF mobilizing regimen, will allow collection of greater than or equal to 5 x 10^6 CD34+ cells/kg in 2 or less apheresis days.

II. To review the timing of intravenous plerixafor administration prior to apheresis and describe our experience.

OUTLINE:

MOBILIZATION: Patients receive cyclophosphamide intravenously (IV). Patients also receive filgrastim subcutaneously (SC) daily beginning approximately 24 hours later.

TREATMENT/APHERESIS: Beginning 10 days after cyclophosphamide, patients receive plerixafor IV over 30 minutes followed by filgrastim SC on each day of apheresis.

Following the collection of an adequate number of stem cells, patients undergo high-dose chemotherapy and autologous stem cell rescue. Patients are followed post-autologous stem cell transplant for engraftment.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Criteria

* Inclusion and exclusion criteria must be re-evaluated prior to dosing with PLERIXAFOR; if the patient does not meet any of these criteria (excluding the hepatic and hematologic criteria) the patient is not eligible to continue unless Genzyme grants a waiver

Inclusion

* Eligible to undergo autologous transplantation
* Diagnosed with multiple myeloma (MM)
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1
* The patient has recovered from all acute toxic effects of prior chemotherapy
* White Blood Count (WBC) > 2.5 x 10^9/L
* Absolute neutrophil count >1.5 x 10^9/L
* Platelet count > 100 x 10^9/L
* Serum creatinine <= 2.5 mg/dl
* Creatinine clearance >= 50 ml/min (measured or calculated)
* Serum glutamic oxaloacetic transaminase (SGOT) < 2 x ULN (Upper Limit of Normal)
* Serum glutamic pyruvic transaminase (SGPT) < 2 x ULN
* Total bilirubin < 2 x ULN
* Left ventricle ejection fraction > 45% [by normal ECHO (Echocardiogram) or MUGA (MUltiple Gated Acquisition) scan]
* FEV1 (forced expiratory volume in 1 second) > 60% of predicted or DLCO (Carbon Monoxide Diffusing Capacity )> 55% of predicted
* No active infection of hepatitis B or C
* Negative for HIV
* Signed informed consent (may be obtained anytime prior to admission for cytoxan)
* Women of child bearing potential agree to use an approved form of contraception

Exclusion

* A co-morbid condition which, in the view of the investigators, renders the patient at high risk from treatment complications
* A residual acute medical condition resulting from prior chemotherapy
* Brain metastases or carcinomatous meningitis
* Acute infection
* Fever (temp > 38 degrees C/100.4 degrees F)
* Positive pregnancy test in female patients
* Lactating females
* Patients of child-bearing potential unwilling to implement adequate birth control
* Prior treatment with Plerixafor
* Prior stem cell transplant, either autologous or allogeneic
* Prior cyclophosphamide priming
* Heart rate < 50 at screening
* Abnormal ECG (electrocardiogram) with a clinically significant rhythm disturbance or conduction abnormality that in the opinion of the investigator warrants exclusion of the subject from the trial
* Patients with congestive heart failure at screening
* History of atrial fibrillation
* Patients who are currently on medication to control cardiac arrhythmias

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To assess the MTD ( maximum tolerated dose) of IV plerixafor when given post cyclophosphamide and GCSF for stem cell priming.Dose limiting toxicity will be defined as any grade 3 or 4 nonhematologic toxicity. | 12 to 18 months
Tolerability and safety of PLERIXAFOR | 6 months post transplant
  Will be summarized in terms of type, severity (by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v4.0), date of onset, duration, reversibility, and attribution.

SECONDARY OUTCOMES:
Frequency of collecting 5 x 10^6 or more CD34+ cells/kg in 2 or less apheresis days | 5 days post apheresis completion
Percentage of plasma cells | 5 days post apheresis
Completion of 100 days post-transplant | 100 days post-transplant
Overall and disease-free survival | 6months and one year post transplant
Time to engraftment | 6 months post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Krishnan, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States